CLINICAL TRIAL: NCT07113639
Title: Effectiveness of High-volume Corticosteroid Injection Diluted With Saline in Subacromial Impingement Syndrome: A Prospective Randomized Trial
Brief Title: Effectiveness of High-Volume Corticosteroid Injection in Shoulder Impingement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, İsa Cüce, Associate Professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-410
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Shoulder Impingement Syndrome
Keywords: shoulder pain; ultrasound; subacromial bursa; injection; different volumes
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Volume Corticosteroid Injection Group (Experimental): US-guided injection of 1 mL triamcinolone acetonide (40 mg), 1 mL 2% lidocaine, and 8 mL normal saline (total volume: 10 mL).
  Interventions: Procedure: Injection
- Low-volume corticosteroid injection (Active Comparator): US-guided injection of 1 mL triamcinolone acetonide (40 mg), 1 mL 2% lidocaine, and 1 mL normal saline (total volume: 3 mL)
  Interventions: Procedure: Injection

INTERVENTIONS:
Procedure: Injection — US-guided subacromial-subdeltoid injection with 1 mL triamcinolone acetonide (40 mg), 1 mL 2% lidocaine, and 8 mL normal saline (10 mL total)
  Arms: High-Volume Corticosteroid Injection Group
Procedure: Injection — US-guided subacromial-subdeltoid injection with 1 mL triamcinolone acetonide (40 mg), 1 mL 2% lidocaine, and 1 mL normal saline (3 mL total)
  Arms: Low-volume corticosteroid injection

SUMMARY:
This study aimed to compare the effectiveness of high-volume versus low-volume ultrasound-guided corticosteroid injections diluted with saline in patients with subacromial impingement syndrome, finding no significant difference in pain or functional outcomes between the two methods.

DETAILED DESCRIPTION:
Subacromial impingement syndrome (SIS) is commonly treated conservatively with corticosteroid (CS) injections into the subacromial bursa, often combined with local anesthetics (LA). Despite widespread use, there remains no consensus regarding the optimal injection technique, volume, or drug formulation. Some studies suggest high-volume injections may provide superior pain relief, while others show no significant difference. To clarify this, a prospective, double-blind, randomized controlled trial was designed to compare the efficacy and safety of high-volume versus low-volume CS injections in patients with SIS.

Material and methods:

This study is a prospective, double-blind, randomized controlled trial. The study procedure was discussed with the patients, and each participant provided written informed consent.

All patients who were admitted to the outpatient clinic with unilateral shoulder pain within the study period, were screened to assess eligibility for the study The following 3-step checklist was completed for an accurate diagnosis of SIS: history of anterolateral arm pain and exacerbation of symptoms upon raising the shoulder to 90° or higher, a combination of the Neer test, Hawkins-Kennedy test, painful-arc test, and infraspinatus muscle test produced at least 2 positive results and confirmation of the diagnosis by an ultrasound (US) evaluation of the affected shoulder.

The same physiatrist (who had 5 years of experience in musculoskeletal US) performed the complete standard US evaluation of the affected shoulder in each patient, according to the EURO-MUSCULUS/USPRM shoulder scanning protocol. All patients also underwent dynamic US evaluation for SIS . A 3-16-mHz linear probe was used in B mode (Samsung HM70A Plus, Seoul, South Korea). For the US diagnosis of SIS, the subacromial-subdeltoid bursa must have been thicker than 2 mm (bursitis) and a sign of impingement must have been seen on the dynamic evaluations. Any pathological abnormalities associated with SIS (tendinosis, partial-thickness rotator cuff tear, etc.) were also noted.

Outcome Measures:

Detailed in the Outcome Measurements section.

Randomization and blinding After baseline assessment, patients were randomly assigned (1:1) to high-volume (H-VCI) or low-volume (L-VCI) corticosteroid injection groups using computer-generated randomization by an independent secretary. A blinded research assistant prepared the injections. Patients and outcome assessors were blinded to group allocation, but the injector was not blinded due to the differing injection volumes.

Interventions Patients in the H-VCI group received 1 mL of 40 mg triamcinolone acetonide (TA), 1 mL of 2% lidocaine, and 8 mL of normal saline mixture (10 mL total). The patients in the L-VCI group received 1 mL of 40 mg TA, 1 mL of 2% lidocaine, and 1 mL of normal saline mixture (3 mL total).

The physiatrist administered all injections following a standard procedure with US . The patient was taken to the operating room and seated in a chair. The affected arm was placed in the modified Crass position, and the injection site was sterilized and draped. The transducer was placed on the anterosuperior aspect of the shoulder to capture the short axis of the supraspinatus tendon. The subacromial-subdeltoid bursa was visualized between the deltoid muscle and the supraspinatus tendon. Using the in-plane technique, a 21G, 38-mm needle was advanced from lateral to medial to reach the subacromial-subdeltoid bursa. After confirming that the needle tip was inside the bursa, the injectate was administered and its distribution appeared.

Injection-related adverse reactions were monitored and recorded over the following 1-2 h prior to discharge. Following the injections, patients were allowed to take paracetamol (and naproxen 750 mg daily if needed) and were asked to note the dosages that they consumed. Patients were instructed not to take analgesics the day before the follow-up appointment, as this could affect the study results.

All patients were trained once by an experienced physical therapist for a home exercise regimen and were then given a leaflet. The regimen consisted of a combination of range of motion, stretching, scapular stabilization, and rotator cuff resistance exercises. Each patient was instructed to begin this exercise program 4 days after the injection.

Data collection and assessment All patients completed standard questionnaires that collected demographic (age, gender, hand dominance, weight, and height) and current shoulder-pain-related data.

The primary outcome measure was the Shoulder Pain and Disability Index (SPADI) score, which evaluates shoulder pain and disability.

Secondary outcomes included Visual Analog Scale (VAS: pain at night, rest, and movement), Western Ontario Rotator Cuff Index Score (WORC) , and active range of motion (AROM: abduction, flexion, internal/external rotation).

All assessments were performed by a blinded researcher. Evaluations were conducted at baseline, 1 hour, 4 weeks, and 12 weeks post-injection. VAS was assessed at all time points; SPADI, WORC, and AROM were assessed at 4 and 12 weeks.

At 4 and 12 weeks, exercise adherence (never, sometimes, always) was also recorded.

Statistical Analysis Sample size was calculated using G*Power (v3.1.9.4) based on a 10-point minimal clinically important difference in SPADI, with a standard deviation of 14, α = 0.05, and power (β) = 80%, requiring 64 patients. To account for 10% attrition, 70 patients were enrolled.

Analyses were performed using SPSS 22.0 (IBM Corp., Armonk, NY, USA). Data were presented as mean ± SD or median (IQR) for continuous variables, and frequency (%) for categorical variables. Normality was assessed using the Shapiro-Wilk test. Independent t-test or Mann-Whitney U test was used for between-group comparisons, and chi-square test for categorical data.

All outcomes were analyzed based on the intention-to-treat principle, with missing data handled via multiple imputation. Within-group changes were analyzed using the Friedman test. Percent changes from baseline to 4 and 12 weeks were calculated and compared between groups. Post-hoc pairwise comparisons were conducted with the Dunn-Bonferroni test. Statistical significance was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of subacromial impingement syndrome (SIS)
* Age over 18 years
* Shoulder pain lasting longer than 4 weeks
* Shoulder pain with a visual analogue scale (VAS) score of 3 or higher
* Passive shoulder range of motion within normal limits

Exclusion Criteria:

* Full-thickness tear or calcification of the rotator cuff in the affected shoulder
* Adhesive capsulitis
* History of trauma or surgery in the affected shoulder
* History of injection into the affected shoulder within the previous 6 months
* History of systemic rheumatic disease, malignancy, or coagulopathy
* Suspected cervical radiculopathy
* History of allergy to local anesthetics (LA) and/or corticosteroids (CS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index score | evaluated at 4 and 12 weeks before injection
  This index assesses shoulder-related pain (5 items) and disability (8 items), for a total of 13 items. Each item is scored from 0 (no pain or difficulty) to 10 (worst pain or very difficult). The score is then converted to a 100-point scale, with higher scores reflecting higher levels of shoulder pain and disability .

SECONDARY OUTCOMES:
Visual Analog Scale (VAS): | before injection, 1 hour later, at 4 and 12 weeks
  A 100-mm horizontal line is used, with the two extremes of the parameter to be assessed labeled at each end. The patient is asked to indicate their perceived condition by marking a point or drawing a line on the scale that best reflects their current state. VAS is commonly employed to numerically document pain intensity as well as the patient's subjective global health assessment.
Western Ontario Rotator Cuff Index Score | evaluated at 4 and 12 weeks before injection
  The WORC consists of 21 items representing five domains (physical symptoms, sports and recreation, work, lifestyle, and emotions). Each item is scored from 0 to 100 (100 mm VAS). The total score, obtained by summing the scores of all items, is expressed as a percentage of normal. A lower percentage reflects a worse quality of life associated with the affected shoulder.
Active Range of Motion | evaluated at 4 and 12 weeks before injection
  active range of motion of the shoulder complex was measured in the supine position using a standard goniometer. These measurements included abduction in the frontal plane, forward flexion, internal rotation, and external rotation with the arm at 90 ° - of abduction.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Faculty of Medicine Hospital, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boonard M, Sumanont S, Arirachakaran A, Apiwatanakul P, Boonrod A, Kanchanatawan W, Kongtharvonskul J. Short-term outcomes of subacromial injection of combined corticosteroid with low-volume compared to high-volume local anesthetic for rotator cuff impingement syndrome: a randomized controlled non-inferiority trial. Eur J Orthop Surg Traumatol. 2018 Aug;28(6):1079-1087. doi: 10.1007/s00590-018-2149-3. Epub 2018 Feb 8. PMID 29423865
- [Result] Sumanont S, Boonard M, Peradhammanon E, Arirachakaran A, Suwankomonkul P, Oungbumrungpan W, Kongtharvonskul J. Comparative outcomes of combined corticosteroid with low volume compared to high volume of local anesthetic in subacromial injection for impingement syndrome: systematic review and meta-analysis of RCTs. Eur J Orthop Surg Traumatol. 2018 Apr;28(3):397-407. doi: 10.1007/s00590-017-2056-z. Epub 2017 Oct 12. PMID 29027006
- [Result] Ge M, Zhang Y, Li Y, Feng C, Tian J, Huang Y, Zhao T. Publication Trends and Hot Spots in Subacromial Impingement Syndrome Research: A Bibliometric Analysis of the Web of Science Core Collection. J Pain Res. 2022 Mar 28;15:837-856. doi: 10.2147/JPR.S348528. eCollection 2022. PMID 35370418